CLINICAL TRIAL: NCT03353493
Title: Neural, Molecular and Psychological Mechanisms and Predictors of Treatment Response to Mindfulness-based Cognitive Therapy in the Treatment of Recurrent Major Depressive Disorder
Brief Title: Mechanisms of Mindfulness-Based Cognitive Therapy in the Treatment of Recurrent Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: University of Oxford (Other); VIA University College (Other); University of York (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Anne Maj van der Velden, PhD fellow, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 314 #2016-051-000001
Record Dates: First submitted 2017-09-08; First posted 2017-11-27 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Major Depressive Disorder, Recurrent
Keywords: Mindfulness-Based Cognitive Therapy; Neural, psychological and molecular mechanisms
MeSH Terms: conditions — Depressive Disorder, Major; Recurrence

STUDY DESIGN:
Intervention Model Description: Randomised to Mindfulness-based cognitive therapy plus treatment as usual, or treatment as usual.
Who Masked: Outcomes Assessor
Masking Description: Participants are masked at baseline assessment to treatment allocation. Outcome assessors are masked to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBCT + TAU (Experimental): Mindfulness-based Cognitive Therapy (MBCT) a 8 week group based intervention delivered according to the protocol by Segal, Williams and Teasdale (2013) plus treatment as usual (TAU) . TAU is restricted to antidepressant medication and no psychological therapy.
  Interventions: Behavioral: MBCT; Other: TAU
- TAU (Other): Treatment as Usual (TAU). TAU is restricted to antidepressant medication and no psychological therapy.
  Interventions: Other: TAU

INTERVENTIONS:
Behavioral: MBCT — Mindfulness-Based Cognitive Therapy (MBCT) is an 8 week manualised group intervention. MBCT will be delivered according to the manual by Segal, Williams & Teasdale (2013).
  Arms: MBCT + TAU
Other: TAU — Treatment as usual (TAU)

SUMMARY:
The primary purpose of this study is to investigate neural mechanisms and predictors of treatment outcome in Mindfulness-Based Cognitive Therapy (MBCT) for recurrent Major Depressive Disorder.

DETAILED DESCRIPTION:
AIM AND HYPOTHESES

The primary aim is to investigate treatment mechanisms of MBCT and markers of relapse risk.

Controlled design:

First, we aim to first investigate the effect of treatment on clinical outcomes in the controlled design post treatment and at 3 months follow up. Second, we will run mediation analyses of hypothesized mechanisms (increased mindfulness skills, decentering, interoceptive and decreased rumination, and change in neural connectivity in a priori networks), and finally check for moderating influences of vulnerability markers (childhood trauma, no. episodes of depression and residual symptoms).

Prospective design:

We aim to investigate predictors of relapse risk at 12 month follow treatment using i) baseline markers and ii) mechanism outcomes that change significantly due to treatment, and iii) check for moderating influences of vulnerability markers

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years
2. Meeting DSM-IV criteria for a history of recurrent Major Depressive Disorder (MDD) with or without a current episode of depression
3. Recurrent MDD evaluated a being the primary disorder.
4. Danish literacy

Exclusion Criteria:

1. A history of schizophrenia, schizoaffective disorder, bipolar disorder, current severe substance abuse, organic mental disorder, current/past psychosis, pervasive developmental delay, persistent antisocial behaviour, persistent self-injury requiring clinical management/therapy
2. Formal concurrent psychotherapy
3. Previous Mindfulness-Based Cognitive Therapy/Mindfulness-Based Stress Reduction
4. Anti-psychotic medication and benzodiazepines
5. Standard exclusion criteria for undergoing magnetic resonance imaging (MRI) procedures for research purposes, i.e., claustrophobia, pregnancy, cardiac pacemaker, prosthetic heart valve, neurostimulator, implanted pumps, cochlear implants, non-MR-compatible implants or devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Change in neural connectivity | Baseline and 8 weeks
  Neural connectivity will be measured with functional magnetic resonance (fMRI). Selected a priory networks for seed-based analyses: Default mode Network and Salience Network

SECONDARY OUTCOMES:
Change in mindfulness skills | Baseline and 8 weeks
  Five Factor Mindfulness Questionnaire (FFMQ)
Change in decentering | Baseline and 8 weeks
  Experiences Questionaire (EQ)
Change in rumination | Baseline and 8 weeks
  Rumination Response Scale (RRS)
Change in emotional processing bias | Baseline and 8 weeks
  Facial Expression Recognition task (FERT)
Change in interoceptive awareness | Baseline and 8 weeks
  Multidimensional Assessment of Interoceptive Awareness (MAIA)
Change in perceived stress | Baseline and 8 weeks
  Perceived Stress Scale (PSS)
Time to relapse or recurrence of depression | 12 months follow up
  Structured clinical interview for DSM-IV
Change in depressive symptoms | Baseline and 8 weeks
  Quick Inventory for Depressive Symptomology (QIDS-SR)
Change in interleukin gene expression | Baseline and 8 weeks
  IL-1, IL-2, IL-4,IL-6, IL-8, IL-10, IL-12p70, IL-13,
Change in interleukin protein expression | Baseline and 8 weeks
  IL-1, IL-2, IL-4,IL-6, IL-8, IL-10, IL-12p70, IL-13,
Change in gene expression of norepinephrine transporter | Baseline and 8 weeks
  Norepinephrine transporter (NET)
Change in gene expression of glutamate receptor | Baseline and 8 weeks
  Glutamate receptor (GRM7)
Change in gene expression of TNF | Baseline and 8 weeks
  Change in gene expression of tumor necrosis factor (previous nomenclature TNF-alfa)
Change in protein expression of tumor necrosis factor | Baseline and 8 weeks
  Tumor necrosis factor
cRP expression | Baseline and 8 weeks
  c reactive protein expression
Change in NF-kB gene expression | Baseline and 8 weeks
  Nuclear factor kappa-light-chain-enhancer of activated B cells gene expression
Change in NF-kB protein expression | Baseline and 8 weeks
  Nuclear factor kappa-light-chain-enhancer of activated B cells protein expression
Change in INFG gene expression | Baseline and 8 weeks
  Interferon gamma gene expresison
Change in Interferon gamma protein expression | Baseline and 8 weeks
  Interferon gamma protein expresison
Mitochondrial DNA Copy Number | Baseline and 8 weeks
  Copy number is assessed using quantitative real-time-PCR

OTHER OUTCOMES:
fMRI BOLD secondary and whole brain analyses | Baseline and 8 weeks
  fMRI BOLD whole brain analyses (data-driven) and secondary subcortical seed-based analyses: As seeds we preselect hippocampus, the amygdala and striatum
Global Gene expression with focus on genes involved in mitochondrial function, the respiratory chain. | Baseline and 8 weeks
  HG-U133 Plus 2.0 GeneChip (Affymetrix)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Maj van der Velden, Msc, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van der Velden AM, Scholl J, Elmholdt EM, Fjorback LO, Harmer CJ, Lazar SW, O'Toole MS, Smallwood J, Roepstorff A, Kuyken W. Mindfulness Training Changes Brain Dynamics During Depressive Rumination: A Randomized Controlled Trial. Biol Psychiatry. 2023 Feb 1;93(3):233-242. doi: 10.1016/j.biopsych.2022.06.038. Epub 2022 Jul 22. PMID 36328822
- See also: Study website — http://interactingminds.au.dk/projects/mindfulness-and-the-prevention-of-depression/